CLINICAL TRIAL: NCT04216524
Title: Phase 2 Clinical Trial for Comprehensive Treatment Program for Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN): Tagraxofusp (SL-401) in Combination With HCVAD/Mini-CVD and VENETOCLAX
Brief Title: Venetoclax, SL-401, and Chemotherapy for the Treatment of Blastic Plasmacytoid Dendritic Cell Neoplasm
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0587; NCI-2019-08358 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0587 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; tagraxofusp; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SL-401, venetoclax, chemotherapy) (Experimental): See detailed description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Prednisone; Biological: Rituximab; Biological: Tagraxofusp-erzs; Drug: Venetoclax; Drug: Vincristine

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, IV, or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Biological: Tagraxofusp-erzs — Given IV
  Other Names: Diphtheria Toxin(388)-Interleukin-3 Fusion Protein; DT(388)-IL3 Fusion Protein; DT388IL3 fusion protein; Elzonris; IL3R-targeting Fusion Protein SL-401; SL-401; Tagraxofusp; Tagraxofusp ERZS
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial studies how well venetoclax, SL-401, and chemotherapy works in treating patients with blastic plasmacytoid dendritic cell neoplasm. Venetoclax may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. SL-401 is a recombinant protein consisting of IL-3 linked to a toxic agent called DT. IL-3 attaches to IL-3 receptors on tumor cells in a targeted way and delivers DT to kill them. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax and SL-401 with chemotherapy may be an effective treatment for patients with blastic plasmacytoid dendritic cell neoplasm.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate progression-free survival (PFS) at 12 months of venetoclax (VEN) in combination with chemotherapy and SL-401 (tagraxofusp [TAG]) in patients with newly diagnosed blastic plasmacytoid dendritic cell neoplasm (BPDCN).

SECONDARY OBJECTIVES:

I. To determine the safety of the SL-401 in combination with VEN and in combination with chemotherapy in patients with newly diagnosed BPDCN by toxicity and futility monitoring.

II. To determine the efficacy by measurement of progression free survival (PFS), overall response rate (ORR): complete response (CR) and complete response with incomplete marrow recovery (CRi), clinical complete response (CRc) and remission duration of SL-401 in combination with chemotherapy and VEN in patients with newly diagnosed BPDCN.

III. To determine the rate of stem cell translant (SCT) within the first 8 cycles (understanding that some patients won't get SCT) in patients with newly diagnosed BPDCN.

EXPLORATORY OBJECTIVES:

I. To examine expression and function of BCL-2 family proteins and its modulation by VEN in BPDCN blasts.

II. To determine the rate of minimal residual disease (MRD) negativity in patients achieving CR/CRi/CRc and its correlation with disease-free survival (DFS) and overall survival (OS).

III. To determine CD123 levels pre- and post-therapy. IV. To determine molecular mutations pre-and post- therapy as part of 81-gene panel by next-generation sequencing.

OUTLINE:

INDUCTION:

CYCLE 1: Patients receive tagraxofusp-erzs (SL-401) intravenously (IV) once daily (QD) over 15 minutes on days 1-5.

CYCLES 2, 4, 6, and 8: Patients receive tagraxofusp-erzs IV QD over 15 minutes on days 1-5, and venetoclax orally (PO) QD on days 1-14 of cycle 2, and days 1-7 of cycles 4, 6, and 8.

CYCLES 3 and 7: Patients receive venetoclax PO QD on days 1-7. Patients whose age < 60 receive hyper-CVAD and age >= 60 receive mini-hyper-CVD. Patients may receive rituximab IV over 90 minutes on days 1 and 8, methotrexate intrathecally (IT) on day 2, and/or cytarabine IT on day 8. Patients also receive venetoclax PO QD on days 1-7.

HYPER-CVAD (AGE < 60): Patients receive cyclophosphamide IV over 3 hours every 12 hours (Q12H) on days 1-3, vincristine IV over 15 minutes on days 1 and 8, dexamethasone orally (PO) or IV over 30 minutes on days 1-4 and 11-14, and doxorubicin IV over 24 hours on day 4.

MINI-HYPER-CVD (AGE >= 60): Patients receive cyclophosphamide IV over 3 hour Q12H on days 1-3, vincristine IV over 15 minutes on days 1 and 8, dexamethasone PO or IV over 30 minutes on days 1-4 and 11-14.

CYCLE 5: Patients receive venetoclax PO QD on days 1-7. Patients who age < 60 receive MTX/AraC and age >= 60 receive mini-MTX/AraC. Patients may receive rituximab IV over 4-6 hours on days 1 and 8, cytarabine IT on day 5, and/or methotrexate IT on day 8.

MTX/ARAC (AGE < 60): Patients receive methotrexate IV over 24 hours on day 1, and cytarabine IV over 3 hours Q12H on days 2 and 3.

MINI-MTX/ARAC (AGE >= 60): Patients receive methotrexate IV over 24 hours on day 1, methylprednisolone IV over 2 hours Q12H on days 1-3, and cytarabine IV over 3 hours Q12H on days 2 and 3.

ALL CYCLES: Treatment repeats every 28 days for 8 cycles in the absence of disease progression and unacceptable toxicity.

MAINTENANCE: Patients receive venetoclax PO QD on days 1-7, POMP chemotherapy during cycles 1-5, 7-11, and 13-17, and SL-401 IV QD on days 1-5 of cycles 6, 12, and 18. Treatment repeats every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity.

POMP: Patients receive mercaptopurine PO three time daily (TID) on days 1-28, vincristine IV over 15 minutes on day 1, prednisone PO QD on days 1-5, and methotrexate PO once weekly.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naïve or relapsed refractory patients with histologically confirmed diagnosis of blastic plasmacytoid dendritic cell neoplasm (BPDCN) per 2016 WHO criteria
2. Front line participants may have received emergent chemotherapy prior to study enrollment:

   1. One prior cycle of SL-401, or other BPDCN-directed therapy, will be allowed prior to entering the study.
   2. Prior or concomitant doses of ARA-C (cytarabine) or Hydroxyurea are allowed on before or during the study for proliferative disease due to BPDCN.
3. Relapsed/refractory participants may have received at least one prior cycle of therapy.
4. Age ≥ 18 years
5. ECOG performance status 0, 1, or 2 (see APPENDIX B)
6. Adequate organ function as defined by:

   * Albumin ≥ 3.2 g/dL (in the absence of receipt of intravenous albumin in the previous 72 hours)
   * Serum creatinine < 1.5x ULN
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN
   * Total bilirubin < 1.5x ULN (if total bilirubin is > 1.5x but < 3x ULN, and thought to be elevated due to Gilbert's disease or the patient's BPDCN, the subject may be eligible but must discuss with the PI)
7. Ability to understand and the willingness to sign a written informed consent document.
8. Able to adhere to study visit schedule and other protocol requirements including follow-up for survival assessment
9. Women of child-bearing potential and men enrolled on this protocol must agree to use adequate contraception for the duration of study participation and for 2 months after completion VEN administration. Acceptable birth control methods allowed to be used while on study include:

   * Birth control pills or injections
   * Intrauterine devices (IUDs)
   * Double-barrier methods for example condom in combination with spermicide. Males should not donate sperm while on study and for at least 8 weeks after the last dose of SL-401.
10. Left ventricular ejection fraction ≥ institutional lower limit of normal by MUGA scan or echocardiogram within 30 days of first protocol treatment.

Exclusion Criteria:

1. Participants is pregnant or breastfeeding
2. Known active hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
3. Major surgery or radiation therapy within 14 days prior to the first study dose
4. Symptomatic or untreated leptomeningeal disease or spinal cord compression
5. Participants with active heart disease (New York Heart Association (NYHA) class 3-4 as assessed by history and physical examination, unstable angina/stroke/myocardial infarction within the last 6 months)
6. Malabsorption syndrome or other conditions that preclude enteral route of administration
7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the participants inappropriate for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 6 years
  The median PFS time will be estimated by Bayesian posterior estimates. Estimated using the Kaplan-Meier method.
Incidence of adverse events | Up to 6 years
  Will be reported by type, frequency and severity. Highest toxicity grades per patient per course will be tabulated for selected adverse events and laboratory measurements.
Overall response rate | Up to 6 years
  Overall response rate along with complete remission and complete remission with incomplete hematologic recovery will be estimated along with 95% confidence interval.
Rate of stem cell transplant | Up to 6 years
  The response rate will be compared between subgroups (e.g. minimal residual disease negativity, etc.) by Fisher's exact test, and Wilcoxon rank test will be used to compare the patient clinical information (e.g., protein expression) between subgroups such as response and non-response.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pemmaraju, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org